CLINICAL TRIAL: NCT02848144
Title: Pediatric Immune Response to Infectious Shock
Acronym: PedIRIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 69HCL16_0478
Record Dates: First submitted 2016-07-21; First posted 2016-07-28 (Estimated); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Severe Pediatric Infectious Shock
Keywords: Immunoparalysis; immune response; sepsis; toxic shock syndrome
MeSH Terms: conditions — Sepsis; Shock, Septic | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Children with infectious shock (Other): Children aged from 1 month to <18 years. In 3 stratified groups : <2 years, 2-8 years, and >8 years. About one third of the patients are expected in each age-group.
  Interventions: Other: blood samples; Other: Collection of nosocomial infections
- Control group: healthy children (Other): Healthy children aged-matched to cases (same stratification group, about 20 per age group); They will be hospitalized for an elective surgery (dental, ENT, maxillofacial, urologic, hernia surgery, neurosurgery without massive hemorrhage) and without any infection.
  Interventions: Other: blood samples; Other: Collection of nosocomial infections

INTERVENTIONS:
Other: blood samples
Other: Collection of nosocomial infections

SUMMARY:
Infectious shocks are associated with high mortality rates (20-40%). Anti-inflammatory strategies based on the postulate that mortality related to sepsis is mainly due to an overwhelming pro-inflammatory immune response have failed. Some patients surviving this initial phase can develop immune dysfunctions because the compensatory mechanisms become deleterious when they persist over time. The persistence of immunosuppression at day 3 or 5 is independently associated with more nosocomial infections and higher mortality rate. The clinical and laboratory evidence for sepsis induced immunosuppression have been recently reviewed by Hotchkiss et al. Apoptosis-induced depletion of immune effector and blood studies from septic patients showed decreased production of pro-inflammatory cytokines, decreased HLA-DR expression, increased percentage of regulatory T cells, and increased production of programmed cell death (PD)-1. Some small positive phase 2 trials of biomarker guided immune enhancing agents granulocyte-macrophage colony stimulating factor (GM-CSF) and interferon γ (IFN γ) have been reported.

There are insufficient data showing that such an immunosuppression exists in children. Only one study performed in children with organ dysfunctions admitted to pediatric intensive care unit (PICU), showed that 34% of them developed immunosuppression. This study was performed on a heterogeneous population and immunological analyses were limited. Therefore, there is a crucial need of studies on septic patients with matched controls to provide more evidence that the same paradigm exists in children. The collaboration of laboratories with a high level of experience in this domain, and a clinical unit with a high potential of recruitment of children with severe infectious shock should allow us to perform the first prospective study specifically done in children with infectious shock.

The main hypothesis is that children with severe infectious shock developed sepsis-induced immunosuppression as shown in adults. This will be assessed by the expression of HLA-DR on monocytes' surface. We make the hypothesis that children who become immunosuppressed are more prone to develop secondary nosocomial infectious and stayed longer in PICU and in hospital.

Children aged from 1 month to 17 years, admitted to PICU at HFME Lyon-Bron are eligible if they have the criteria for severe sepsis or septic shock, defined by the "Surviving Sepsis Campaign 2012" or those of Toxic Shock Syndrome (TSS) (definitions of CDC - Center for Disease Control). An information leaflet will be issued to parents and children / adolescents and they will be informed of their right to object to the search. Are provided as part of this research:

* Immunological measures (mHLA -DR) in three stages: in the first 48 hours, between D3/5 and D7/9. The volume of collected blood will not exceed 2.4 ml / kg.
* The collection of nosocomial infections and status at D30 A control group of patients hospitalized for surgery without sepsis or toxic shock criteria will be recruited in the same hospital by ICU investigators and matched for age. Similarly controls will be given oral and written information and they will have the opportunity to deny inclusion. They will have the same exams as the first group of patients.

ELIGIBILITY:
Inclusion Criteria Infectious shock group:

* Children aged from 1 month to <18 years
* Diagnosis of severe infectious shock at PICU or within the first 24 hours following PICU admission: severe sepsis or septic shock, defined by Surviving Sepsis Campaign 2012, or Toxic Shock Syndrome, defined by CDC criteria.

Inclusion Criteria Control group:

* Healthy children aged matched to cases
* Hospitalized for an elective surgery (dental, ENT, maxillofacial, urologic, hernia surgery, neurosurgery without massive hemorrhage)
* Without any criteria of infection.

Exclusion Criteria (both groups):

* Chronic inflammatory disease;
* Immunodeficiency;
* Long-term corticosteroids;
* Ongoing immunosuppressive treatment;
* Transplanted patients;
* Tumors, hematological diseases;
* No health insurance coverage;
* Refusal to participate (from parents and/or patient) or inability to understand information.

Ages: 1 Month to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 105 (Actual)
Dates: Start 2014-09-26 (Actual); Primary Completion 2018-08-04 (Actual); Study Completion 2018-08-04 (Actual)

PRIMARY OUTCOMES:
proportion of patients with a mHLA-DR level <30% | up to Day 9
  mHLA-DR is measured by flow cytometry
proportion of patients with a mHLA-DR level significantly lower than healthy children. | in the pre-operative period
  mHLA-DR is measured by flow cytometry

SECONDARY OUTCOMES:
total lymphocytes | Day 1
  From the whole blood samples, each lymphocytes sub-populations are determined by flow-cytometry with addition of specific monoclonal antibodies
total lymphocytes | between Day 3 and day 5
  From the whole blood samples, each lymphocytes sub-populations are determined by flow-cytometry with addition of specific monoclonal antibodies
total lymphocytes | between Day 7 and day 9
  From the whole blood samples, each lymphocytes sub-populations are determined by flow-cytometry with addition of specific monoclonal antibodies
levels of CD4+ | Day 1
  From the whole blood samples, each lymphocytes sub-populations are determined by flow-cytometry with addition of specific monoclonal antibodies
levels of CD4+ | between Day 3 and day 5
  From the whole blood samples, each lymphocytes sub-populations are determined by flow-cytometry with addition of specific monoclonal antibodies
levels of CD4+ | between Day 7 and day 9
  From the whole blood samples, each lymphocytes sub-populations are determined by flow-cytometry with addition of specific monoclonal antibodies
levels of CD25+ | day 1
  From the whole blood samples, each lymphocytes sub-populations are determined by flow-cytometry with addition of specific monoclonal antibodies
levels of CD25+ | between Day 3 and day 5
  From the whole blood samples, each lymphocytes sub-populations are determined by flow-cytometry with addition of specific monoclonal antibodies
levels of CD25+ | between Day 7 and day 9
  From the whole blood samples, each lymphocytes sub-populations are determined by flow-cytometry with addition of specific monoclonal antibodies
levels of T lymphocytes (Treg) | Day 1
  From the whole blood samples, each lymphocytes sub-populations are determined by flow-cytometry with addition of specific monoclonal antibodies
levels of T lymphocytes (Treg) | between Day 3 and day 5
  From the whole blood samples, each lymphocytes sub-populations are determined by flow-cytometry with addition of specific monoclonal antibodies
levels of T lymphocytes (Treg) | between Day 7 and day 9
  From the whole blood samples, each lymphocytes sub-populations are determined by flow-cytometry with addition of specific monoclonal antibodies
dosage of cytokines | Day 1
dosage of cytokines | between Day 3 and day 5
dosage of cytokines | between Day 7 and day 9
Number of nosocomial infections | up to Day 30
Type of nosocomial infections | up to Day 30
  bacteremia, ventilator-associated pneumonia, urinary tract infection, other sites.
Mortality | up to Day 30
Length of vasoactive treatments | up to Day 30

CONTACTS AND LOCATIONS:
Overall Officials: Etienne JAVOUHEY, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hospices Civils de Lyon, Lyon, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Remy S, Kolev-Descamps K, Gossez M, Venet F, Demaret J, Javouhey E, Monneret G. Occurrence of marked sepsis-induced immunosuppression in pediatric septic shock: a pilot study. Ann Intensive Care. 2018 Mar 13;8(1):36. doi: 10.1186/s13613-018-0382-x. PMID 29536210